CLINICAL TRIAL: NCT04413513
Title: A Pilot Study on Randomized Control Trial Comparing Integrated Attention Training Program (IATP) and Health Education on Preservation of Cognitive Functioning in Chinese Older Adults With Anxiety Symptoms.
Brief Title: Effect of IATP on Cognitive Functioning in Anxious Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ada Wai Tung FUNG, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-BE11
Record Dates: First submitted 2018-08-13; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Anxiety Symptoms
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Attention Training Program (Experimental): The intervention group (I) will receive "integrated attention training program (IATP)" on a variety of structured attention tasks by an intervention instructor. It is considered to be simple and safe but effective enough for cognitive health promotion.
  Interventions: Other: Integrated Attention Training Program (IATP)
- Health Education (Placebo Comparator): The control group (C) will receive health educational sessions on health concerns and physical diseases commonly found in old age during the invention period.
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Integrated Attention Training Program (IATP) — Integrated attention training program (IATP) is a newly developed cognitive training programs that combined relaxation technique with integrated attentional training into daily life activity.
  Arms: Integrated Attention Training Program
Other: Health Education — Health educational sessions on health concerns and physical diseases commonly found in old age
  Arms: Health Education

SUMMARY:
Older adults with anxiety symptoms was found to be associated with greater risk of dementia. Interventions targeting signs as early as in the pre-symptomatic phase could be most effective in early prevention of dementia. On reviewing the identified non-pharmacological interventions, integrated attention training program (IATP) is proposed to target older adults with anxiety symptoms in Hong Kong.

DETAILED DESCRIPTION:
Older adults with anxiety disorders or symptoms are not in the consideration of management for dementia prevention. However, the condition is found to be associated with profound negative subsequent decline on both functioning and cognition. While epidemiological studies reported high prevalence in older population, its symptoms are often overlooked in the presence of other age-related diseases in the community as well as among the health professionals. It is expected that cognitive and functional disabilities secondary to this condition will pose a significant burden to the existing healthcare system. Therefore, targeting anxious older adults for early intervention may help to cut healthcare costs and to ensure proactive dementia prevention in the long run. The current proposed intervention intends to attenuate the trajectory of cognitive decline at a very early stage and enhance existing cognitive function to delay the onset of dementia.

This study aims to explore whether the use of integrated attention training program (IATP) could improve cognitive performance and functioning in older adults with anxiety symptoms. In particulars, we aim

1. To examine the cognitive effect of 4 week integrated attention training program (I) and health education (C) in older adults with anxiety symptoms.
2. To examine the 4 week integrated attention training program (I) and health education (C) in alleviating mood symptoms in older adults with anxiety symptoms.
3. To examine the acceptability and adherence of the proposed intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged 60 - 90 years; and
2. Presence of subjective memory complaints as measured by memory inventory for the Chinese; and
3. Anxiety symptoms as measured by Hamilton Anxiety Scale (HAM-A) with a score of 18 or above (indicated as mild anxiety symptoms).

Exclusion Criteria:

1. DSM-5 diagnosis of either Major Neurocognitive Disorder due to AD, or Major Vascular Neurocognitive Disorder with small vessel disease. This would include satisfying criteria for significant cognitive decline in at least one of six areas of cognition (memory, perceptual-motor, complex attention, language, executive function and social cognition), and with clinical or neuroimaging features indicative of either AD or small vessel disease; or;
2. Clinical dementia rating larger than or equal to 0.5; or
3. Clinically depressed as assessed by Hamilton Depression Rating Scale with a score of 20 or higher; or
4. Past history of major depressive episode, bipolar affective disorders or psychosis; or
5. Physical frailty that may affect attendance to training sessions; or
6. Currently on psychotropic or other medications know to affect cognition (e.g., benzodiazepines, anti-dementia medication, etc.); or
7. Participants in other cognitive training or intervention for brain health during the study period; or
8. Presence of major neurological deficit including history of stroke, transient ischemic attack or traumatic brain injury; or
9. Significant communicative impairment.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Attention network test (ANT) | T1: baseline, T2: 4th week, T3:12th week
  ANT will measure the changes in attention from baseline to endpoint between the intervention and control groups. Performance was based on (i) accuracy refers to the degree of correctness and also to quality control, which means that if the participant's accuracy fell below 70%, the case would be considered unqualified. (2) reaction time refers to the processing speed. Median values of RT will be used as raw scores to avoid the influence of outliers. The indices will be served to compare the effect of IATP and health education.

SECONDARY OUTCOMES:
Subjective memory complaints (SMC) | T1: baseline, T2: 4th week, T3:12th week
  SMC will be measured by Memory Inventory for the Chinese (MIC-27). It is locally validated among older people with mild cognitive impairment (MCI) and mild dementia. Participants with a positive answer to any of the 27 questions will be categorized as having SCC at baseline. The total score ranges from 0 to 27, with higher marks indicating poor self-efficacy in memory. There is no cut-off for this outcome measure.
Clinical Dementia Rating (CDR) | T1: baseline, T2: 4th week, T3:12th week
  CDR is a semi-structured clinical interview for the severity of cognitive impairment rated along six dimensions of cognition and function, including memory, orientation, judgement and problem solving, community affairs, home, hobbies and personal cares. Scores in each dimension are combined to form a global rating ranging from 0 (not demented), 0.5 (questionable), 1 (mild), 2 (moderate) to 3 (severe dementia). It has been demonstrated that CDR sum of boxes is sensitive to capture early functional changes in the preclinical phase of AD (CDR 0.5)
Digit and visual spans | T1: baseline, T2: 4th week, T3:12th week
  Digit span is a test of attention and verbal working memory. Participants are asked to repeat back a series of digits immediately after presentation, in ascending order starting from 3 and up to 8 digits (i.e., forward), and in reverse order beginning from 2 to 8 digits (i.e., backward). Both trials of each span length are administered until failure on both trials of a span length is obtained.
  Visual span is a test of attention and visual working memory. It measures the ability to reproduce the spatial pattern of tapping sequences on an array of blocks beginning with 2 and going up to 8 blocks plus the ability to reverse the spatial block tapping sequence from 2 up to 7 blocks. Similar to digit span test, both trails of a span length are given until the length reached at which both are failed.
  Changes in digit and visual spans from baseline to endpoint between groups will be served to compare the effect of IATP and health education on executive function
Delayed recall | T1: baseline, T2: 4th week, T3:12th week
  Changes in delayed recall from baseline to endpoint between the intervention and control groups will be served to compare the effect of IATP and health education on episodic memory.
Category verbal fluency tests | T1: baseline, T2: 4th week, T3:12th week
  Category verbal fluency test (CVFT) is test of semantic fluency and executive function. Participants were asked to generate as many exemplars as possible for each of the three semantic categories, namely animals, fruits, and vegetables, in 60 seconds. Their responses were recorded in serial order. Analysis of scoring is based on the total number of words that the participant is able to produce across all three categories. Also, the number of repetitions and intrusions were recorde. Changes in category verbal fluency test from baseline to endpoint between the intervention and control groups were served to compare the effect of IATP and health education on verbal memory.
Trail making tests | T1: baseline, T2: 4th week, T3:12th week
  Chinese trail making test (A and B) is a test providing information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. There are two parts to the Chinese trail test: A, in which the subject needs to connect the Arabic numbers in sequential order, and B, in which the subject alternates between Arabic and Chinese numbers to suit the literacy of local older population. The completion time (in second) and the numbers of errors made during the test are recorded.
  Changes in trail making test from baseline to endpoint between the intervention and control groups will be served to compare the effect of IATP and health education on executive function and processing speed.
Hong Kong - Montreal Cognitive Assessment | T1: baseline, T2: 4th week, T3:12th week
  Changes in Hong Kong - Montreal Cognitive Assessment (HK-MoCA) from baseline to endpoint between the intervention and control groups will be served to compare the effect of IATP and health education on global cognition. The score ranges from 0-30. A HK-MoCA score of 26 or above, which has been used as a cut-off for mild cognitive impairment (MCI) in older people aged 65 or above with more than 10 years of education
The Chinese Neuropsychiatric Inventory (CNPI) | T1: baseline, T2: 4th week, T3:12th week
  The Chinese Neuropsychiatric Inventory (CNPI) would be used to assess changes in 12 neuropsychiatric symptoms. The frequency of each symptom is rated on a scale of 1 (occasionally) to 4 (very frequently). The severity of each symptom is also rated on a scale of 1 to 3. The total score for each domain is calculated by multiplying the frequency by the severity. A total score is calculated by adding all the domain scores together. Higher score indicating more neuropsychiatric disturbances, In the current proposal, CNPI would evaluate potential mood and behavioral changes.
Hamilton Anxiety Scale (HAM-A) | T1: baseline, T2: 4th week, T3:12th week
  Hamilton Anxiety Scale (HAM-A). It will be used to evaluate anxiety symptoms from baseline to endpoint in both groups. It consists of 14 items on different anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where 17 or less indicates mild severity, 18-24 indicates mild to moderate severity and 25-30 moderate to severe.
Hamilton Depression Scale (HAM-D) | T1: baseline, T2: 4th week, T3:12th week
  Hamilton Depression Scale (HAM-D). It is a commonly used scale to evaluate depressive symptoms. It consists of 17 items on different depressive symptoms, a score of 20 and higher is considered as moderate depression.
The Disability Assessment for Dementia (DAD) | T1: baseline, T2: 4th week, T3:12th week
  The Disability Assessment for Dementia (DAD) captures the ability of a subject to perform everyday tasks appropriate for the older community. It assesses functional abilities in both basic and instrumental activities of daily living.It measures different dimensions (expressed in 0-100%) of task performance, including initiation, planning and organization, and effectiveness. Changes in each dimension of the activities of daily living (ADL) were evaluated to compare the effect of IATP and health education on daily functioning.
Lifestyle activity participation questionnaire | T1: baseline, T2: 4th week, T3:12th week
  Lifestyle activities were categorized into four different types: (i) physical exercises (including mind body exercise and strenuous exercise); (ii) cognitive activity; (iii) social activity; and (iv) recreational activity. The total number of activities engaged was counted for each category. Frequency of lifestyle activity participation was defined as the number of times the participants had engaged at a specified interval in the past year: (i) daily; (ii) several times a week; (iii) weekly; (iv) several times a month; (v) monthly; (vi) bimonthly; and (vii) 3 months or longer. Lifestyle activity participation to measure the change of activity pattern before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tung Fung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No